CLINICAL TRIAL: NCT04555278
Title: Repetitive Transcranial Magnetic Stimulation Alone and in Combination With Motor Control Exercise for the Treatment of Patients With Chronic Non-specific Low Back Pain (ExTraStim Trial): Study Protocol for a Randomized Controlled Trial
Brief Title: Combining Non-invasive Brain Stimulation and Exercise to Treat Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hugo Massé-Alarie (Other)
Collaborators: Pfizer (Industry); The Canadian Pain Society (Other); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Hugo Massé-Alarie, Associate Professor, Medicine Faculty, Department of Rehabilitation, Laval University
Organization: Laval University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020-1844
Record Dates: First submitted 2020-09-14; First posted 2020-09-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Chronic Low-back Pain
Keywords: Transcranial Magnetic Stimulation; Motor Control Exercises; Randomized Controlled Trial
MeSH Terms: interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Pseudo-factorial design (rTMS: Active/Sham | Exercises: Yes/No)
Who Masked: Outcomes Assessor
Masking Description: Participants will be masked to rTMS intervention (real or sham) but cannot be blinded to the exercise intervention. However, participants will not be aware of the study design (other arms).
  Therapist delivering the exercise intervention will be masked to rTMS intervention (active vs. sham) but cannot be blinded to exercise intervention (yes vs. no).
  Experimenter delivering the rTMS intervention will be masked to exercise intervention but not to rTMS intervention (real or sham).
  Outcomes assessor will be completely masked to all interventions as all outcomes are questionnaires that will be completed online. Data will be de-identified and the data analyst will be masked to participants and group allocation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active rTMS + Motor control exercises (Experimental): Active (real) repetitive transcranial magnetic stimulation (20 minutes), immediately followed by a session of motor control exercises taught and supervised by a physiotherapist (30 minutes).
  Interventions: Device: Active rTMS; Other: Motor Control Exercises
- Sham rTMS + Motor control exercises (Sham Comparator): Sham repetitive transcranial magnetic stimulation (20 minutes), immediately followed by a session of motor control exercises taught and supervised by a physiotherapist (30 minutes).
  Interventions: Device: Sham rTMS; Other: Motor Control Exercises
- Active rTMS (Experimental): Active (real) repetitive transcranial magnetic stimulation (20 minutes).
  Interventions: Device: Active rTMS
- Sham rTMS (Sham Comparator): Sham repetitive transcranial magnetic stimulation (20 minutes).
  Interventions: Device: Sham rTMS

INTERVENTIONS:
Device: Active rTMS — A figure-of-8 coil connected to a biphasic Magstim Rapid 2 stimulator (The MagstimCo, Whitland, UK) will be used. Coil orientation and position will be guided throughout the experiment by a neuronavigation system (Brainsight, Rogue research, Montreal, QC, Canada). The intensity of rTMS will be set at 95 % of the first dorsal interosseous (FDI) resting motor threshold (RMT).
  Active rTMS will consist of 40 trains of 5 seconds each at 10 Hz (25-s intertrain interval) applied over M1 (on FDI cortical representation), for a total of 2000 stimulations lasting 20 minutes.
  Other Names: Repetitive Transcranial Magnetic Stimulation
  Arms: Active rTMS; Active rTMS + Motor control exercises
Device: Sham rTMS — A sham coil will be use (e.g. equipped with a magnetic shield that blocks the magnetic field). The sham stimulation will last the same duration as the active rTMS (30 min).
  Other Names: Sham Repetitive Transcranial Magnetic Stimulation
  Arms: Sham rTMS; Sham rTMS + Motor control exercises
Other: Motor Control Exercises — The rehabilitation program will consist of a 30-minute session of motor control exercises following the rTMS (Active or Sham) intervention. This approach aims to improve spine health through the optimization of spine loading. The first session will be preceded by an individualized evaluation of the participant's abilities and deficiencies to tailor the training program to each participant.
  Arms: Active rTMS + Motor control exercises; Sham rTMS + Motor control exercises

SUMMARY:
The aim of this study is to evaluate the efficacy of repetitive transcranial magnetic stimulation alone and in combination with motor control exercises on pain and disability for patients with chronic non-specific low back pain.

ELIGIBILITY:
Inclusion Criteria:

* chronic low back pain, defined as "pain in the low back area with or without leg pain above the knee limiting activities or daily routine which has been present for more than 3 months";
* a minimal average pain intensity of 3 out of 10 during the preceding week on a pain numerical rating scale;
* a minimal score of 10 points on the Oswestry disability index (ODI).

Exclusion Criteria:

* specific spinal pathology (fracture, tumor, radiculopathy, spinal infection, etc.);
* a history of back surgery;
* a major orthopedic, neurological, cardiovascular or psychiatric illness;
* low back pain is not the main pain complaint;
* currently using an exercise program to treat their LBP;
* presenting with any specific TMS/rTMS-related exclusion criteria such as previous seizure/convulsion, cochlear implant, specific medication and pregnancy;
* previous use of repetitive transcranial magnetic stimulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Pain intensity (average pain over the last week) | Change from baseline to 4 weeks, 8 weeks, 12 weeks and 24 weeks
  Pain score on a 11-point pain numerical rating scale (PNRS) ranging from 0 to 10, with 0 meaning no pain and 10 the worst pain imaginable.

SECONDARY OUTCOMES:
Disability (ODI) | Change from baseline to 4 weeks, 8 weeks, 12 weeks and 24 weeks
  The Oswestry Disability Index (ODI) version 2.1 is a self-completed questionnaire giving a subjective percentage score of disability. Includes 10 questions rated on a 6-item scale, from 0 to 5 points. The total score ranges from "0" (No disability) to "100" (Maximal disability).
Tampa scale of kinesiophobia (TSK) | Change from baseline to 8 weeks, 12 weeks and 24 weeks
  TSK is used to assess pain-related fear of movement with a 17-item questionnaire. Each item is scored on a 4-point Likert scale. Total score ranges from 17 (minimal pain-related fear of movement) to 58 (maximal pain-related fear of movement).
Global rating of change | Change from baseline to 8 weeks
  A 11-point scale ranging from -5 to 5, to evaluate the perceived change of health status after the intervention.

OTHER OUTCOMES:
Brain imaging using MRI metrics | Baseline
  Resting-state fMRI and diffusion MRI imaging will be acquired on a 3T Philips Scanner (Achieva 3.0T (TX), Philips Healthcare Medical Systems, Best, Netherlands) with an 15-channel head coil.
  Functional and anatomic connection will be assessed between several regions of interest including: the primary motor cortex and the thalamus, the thalamus and the periaqueductal gray, the nucleus accumbens and the medial prefrontal cortex, the uncinate fasciculus.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Massé-Alarie, PhD, Principal Investigator — Laval University
Locations (1):
- CIRRIS (Centre Interdisciplinaire de Recherche en Réadaptation et Intégration Sociale), Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Patricio P, Tittley J, Lucas de Oliveira FC, Roy M, Fakhry N, Macedo LG, Hodges PW, Leonard G, Roy JS, Masse-Alarie H. Repetitive Transcranial Magnetic Stimulation and Motor Control Exercise for Chronic Low Back Pain: The ExTraStim Randomized Placebo-Controlled Trial. J Orthop Sports Phys Ther. 2026 Jan;56(1):1-10. doi: 10.2519/jospt.2025.13681. PMID 41385357
- [Derived] Patricio P, Roy JS, Macedo L, Roy M, Leonard G, Hodges P, Masse-Alarie H. Repetitive transcranial magnetic stimulation alone and in combination with motor control exercise for the treatment of individuals with chronic non-specific low back pain (ExTraStim trial): study protocol for a randomised controlled trial. BMJ Open. 2021 Mar 24;11(3):e045504. doi: 10.1136/bmjopen-2020-045504. PMID 33762244